CLINICAL TRIAL: NCT00094159
Title: Phase I Open-Label, Multicenter, Dose-Escalation Clinical Study of the Safety and Pharmacokinetic Profiles of Weekly Intravenous Administrations of SNS-595 in Patients With Advanced Malignancies
Brief Title: Safety Assessment of Weekly Intravenous Infusions of SNS-595 for the Treatment of Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0002
Record Dates: First submitted 2004-10-14; First posted 2004-10-15 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — vosaroxin

INTERVENTIONS:
Drug: SNS-595

SUMMARY:
The purpose of this study is to determine whether SNS-595 given intravenously weekly for 3 weeks is safe.

DETAILED DESCRIPTION:
Other objectives of this study include measuring pharmacokinetics (how long the drug can be measured in the blood) and determining the dose and dose schedule for the next phase of studies with SNS-595.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent
* 18 years of age
* Advanced solid malignant tumors
* Tumor can be measured and evaluated
* Blood tests are within standard limits
* Normal blood coagulation
* ECOG Performance Status equal to 0 or 1
* Hemoglobin > or = to 9.0 g/dL
* Absolute Neutrophil Count > or = to 1,500
* Platelets > or = to 100,000
* Calculated or measured creatinine clearance < 50 mL/min
* Serum creatinine < or = 1.5 times the upper limit of normal (ULN)
* AST, ALT, Alkaline Phosphatase < 3 times ULN except if there is hepatic involvement then AST, ALT, and Alkaline Phosphatase < or = to 5 times ULN
* Total Bilirubin < or = to 2 mg/dL

Exclusion Criteria:

* Prior exposure to SNS-595
* Pregnant or breastfeeding.
* Women of childbearing potential unwilling to use an approved, effective means of contraception according to the institution's standards.
* Heart attack, stroke/TIA or other blood clotting event (deep vein thrombosis or pulmonary embolus) within 6 months before the screen visit.
* Requires kidney dialysis (hemodialysis or peritoneal).
* Known bleeding disorder (i.e., hemophilia, von Willebrand Disease, coagulopathy, etc.).
* Received an investigational agent or prior chemotherapy or immunotherapy within 28 days before first dose of SNS-595
* Receiving therapeutic anticoagulation therapy (coumadin, heparin, etc.).
* Currently receiving corticosteroids (inhaled steroids for breathing diseases are allowed) or seizure medications.
* Any medical, psychological, or social condition that, in the opinion of the Principal Investigator, would contraindicate the patient's participation in the clinical trial due to safety and or compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Adelman, MD, Study Director — Sunesis Pharmaceuticals
Locations (4):
- United States (4):
  - Arizona Cancer Center, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Stanford University Medical Center, Stanford, California
  - Duke University Medical Center, Durham, North Carolina